CLINICAL TRIAL: NCT03915678
Title: Atezolizumab Combined With BDB001 AnD Immunogenic Radiotherapy in Patients With Advanced Solid Tumors
Acronym: AGADIR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Bergonié (Other)
Collaborators: Roche Pharma AG (Industry); National Cancer Institute, France (Other Government); Eikon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB 2019-01; 2019-000850-78 (EudraCT Number)
Record Dates: First submitted 2019-04-08; First posted 2019-04-16 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor, Adult; Pancreatic Cancer; Virus-associated Tumors; Non Small Cell Lung Cancer; Melanoma; Bladder Cancer; Triple Negative Breast Cancer
Keywords: Immunotherapy; Radiotherapy; Oncology; Metastatic
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Melanoma; Urinary Bladder Neoplasms; Triple Negative Breast Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — BDB001

STUDY DESIGN:
Intervention Model Description: 6 independent single-arm, multicenter, phase II trials, based on 2-stage Simon's optimal design (Simon R, Controlled Clinical Trials 1989):
  * Population 1: pancreatic cancer
  * Population 2: virus-associated tumors
  * Population 3: non-small lung cancer
  * Population 4: soft-tissue sarcoma
  * Population 5: bladder cancer
  * Population 6: triple negative breast cancer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Population 1: Pancreatic cancer (Experimental): Participants with pancreatic cancer will be treated with Atezolizumab combined with BDB001 and radiotherapy.
  Interventions: Drug: Association atezolizumab + BDB001 + RT
- Population 2: Virus-associated tumors (Experimental): Participants with virus-associated tumors will be treated with Atezolizumab combined with BDB001 and radiotherapy.
  Interventions: Drug: Association atezolizumab + BDB001+ RT
- Population 3: anti-PD-1/L1 refractory non-small lung cancer (Experimental): Participants with anti-PD-1/L1 refractory non-small lung cancer will be treated with Atezolizumab combined with BDB001 and radiotherapy.
  Interventions: Drug: Association atezolizumab + BDB001+ RT
- Population 4: Soft-tissue sarcoma (Experimental): Participants with soft-tissue sarcoma will be treated with Atezolizumab combined with BDB001 and radiotherapy.
  Interventions: Drug: Association atezolizumab + BDB001 + RT
- Population 5: anti-PD-1/L1 refractory bladder cancer (Experimental): Participants with anti-PD-1/L1 refractory bladder cancer will be treated with Atezolizumab combined with BDB001 and radiotherapy.
  Interventions: Drug: Association atezolizumab + BDB001 + RT
- Population 6: Triple negative breast cancer (Experimental): Participants with triple negative breast cancer will be treated with Atezolizumab combined with BDB001 and radiotherapy.
  Interventions: Drug: Association atezolizumab + BDB001 + RT

INTERVENTIONS:
Drug: Association atezolizumab + BDB001 + RT — A treatment cycle consits of 3 weeks. Atezolizumab will be administered as a 1-hour infusion on day 1 every 3 weeks (1200 mg).
  BDB001 will be administered by a 30-minute intravenous infusion before atezolizumab, on Days 1, 8, and 15 of cycles 1, 2, and 3. Then from cycle 4 BDB001 will be administered on Day 1 every 3 weeks.
  Radiotherapy will start at least one week after the first administration of atezolizumab and at the latest before the 2nd administration. All participants will be treated by high dose irradiation in stereotactic conditions on non-injected metastasis: 3 to 5 fractions for a total dose between 27 Gy and 60 Gy.
  Arms: Population 1: Pancreatic cancer
Drug: Association atezolizumab + BDB001+ RT — A treatment cycle consits of 3 weeks. Atezolizumab will be administered as a 1-hour infusion on day 1 every 3 weeks (1200 mg).
  BDB001 will be administered by a 30-minute intravenous infusion before atezolizumab, on Days 1, 8, and 15 of cycles 1, 2, and 3. Then from cycle 4 BDB001 will be administered on Day 1 every 3 weeks.
  Radiotherapy will start at least one week after the first administration of atezolizumab and at the latest before the 2nd administration. All participants will be treated by high dose irradiation in stereotactic conditions on non-injected metastasis: 3 to 5 fractions for a total dose between 27 Gy and 60 Gy.
  Arms: Population 2: Virus-associated tumors
Drug: Association atezolizumab + BDB001+ RT — A treatment cycle consits of 3 weeks. Atezolizumab will be administered as a 1-hour infusion on day 1 every 3 weeks (1200 mg).
  BDB001 will be administered by a 30-minute intravenous infusion before atezolizumab, on Days 1, 8, and 15 of cycles 1, 2, and 3. Then from cycle 4 BDB001 will be administered on Day 1 every 3 weeks.
  Radiotherapy will start at least one week after the first administration of atezolizumab and at the latest before the 2nd administration. All participants will be treated by high dose irradiation in stereotactic conditions on non-injected metastasis: 3 to 5 fractions for a total dose between 27 Gy and 60 Gy.
  Arms: Population 3: anti-PD-1/L1 refractory non-small lung cancer
Drug: Association atezolizumab + BDB001 + RT — A treatment cycle consits of 3 weeks. Atezolizumab will be administered as a 1-hour infusion on day 1 every 3 weeks (1200 mg).
  BDB001 will be administered by a 30-minute intravenous infusion before atezolizumab, on Days 1, 8, and 15 of cycles 1, 2, and 3. Then from cycle 4 BDB001 will be administered on Day 1 every 3 weeks.
  Radiotherapy will start at least one week after the first administration of atezolizumab and at the latest before the 2nd administration. All participants will be treated by high dose irradiation in stereotactic conditions on non-injected metastasis: 3 to 5 fractions for a total dose between 27 Gy and 60 Gy.
  Arms: Population 4: Soft-tissue sarcoma
Drug: Association atezolizumab + BDB001 + RT — A treatment cycle consits of 3 weeks. Atezolizumab will be administered as a 1-hour infusion on day 1 every 3 weeks (1200 mg).
  BDB001 will be administered by a 30-minute intravenous infusion before atezolizumab, on Days 1, 8, and 15 of cycles 1, 2, and 3. Then from cycle 4 BDB001 will be administered on Day 1 every 3 weeks.
  Radiotherapy will start at least one week after the first administration of atezolizumab and at the latest before the 2nd administration. All participants will be treated by high dose irradiation in stereotactic conditions on non-injected metastasis: 3 to 5 fractions for a total dose between 27 Gy and 60 Gy.
  Arms: Population 5: anti-PD-1/L1 refractory bladder cancer
Drug: Association atezolizumab + BDB001 + RT — A treatment cycle consits of 3 weeks. Atezolizumab will be administered as a 1-hour infusion on day 1 every 3 weeks (1200 mg).
  BDB001 will be administered by a 30-minute intravenous infusion before atezolizumab, on Days 1, 8, and 15 of cycles 1, 2, and 3. Then from cycle 4 BDB001 will be administered on Day 1 every 3 weeks.
  Radiotherapy will start at least one week after the first administration of atezolizumab and at the latest before the 2nd administration. All participants will be treated by high dose irradiation in stereotactic conditions on non-injected metastasis: 3 to 5 fractions for a total dose between 27 Gy and 60 Gy.
  Arms: Population 6: Triple negative breast cancer

SUMMARY:
Basket trial concept to independently and simultaneously assess the effects of the association of atezolizumab + BDB001 + radiotherapy in multiple solid tumors.

DETAILED DESCRIPTION:
6 independent, multicenter, prospective, single-arm phase II trials, based on 2-stage Simon's optimal design, will be conducted in parallel to assess the efficacy of atezolimab + BDB001+ radiotherapy, separately, in distinct populations of solid tumors:

* Population 1: pancreatic cancer
* Population 2: virus-associated tumors
* Population 3: anti-PD-1/L1 refractory non-small lung cancer
* Population 4: soft-tissue sarcoma
* Population 5: anti-PD-1/L1 refractory bladder cancer
* Population 6: triple negative breast cancer

ELIGIBILITY:
Inclusion criteria:

1. histologically confirmed pancreatic cancer, virus-associated tumors [including papillomaviruses-related cancers (cervical, head and neck, and nasal), Epstein-Barr virus (nasopharyngeal carcinoma) and Kaposi's sarcoma-associated herpes virus), non-small cell lung cancer, soft-tissue sarcomas, bladder cancer, triple negative breast cancer. For population 4, diagnosis must be confirmed by the RRePS Network as recommended by the French NCI. For population 2, papillomavirus-related cancers must be eligible whatever the genotype but in case of viral genotype is not available, IHC p16 positive must be provided, hepatocellular carcinoma must be confirmed by Hepatite B or C infection, HHV-8 and Epstein-Barr virus related cancers must be confirmed by molecular analysis,
2. Metastatic disease,
3. Age ≥ 18 years,
4. ECOG ≤ 1,
5. At least two lesions: one extra cerebral lesion that can be treated by radiotherapy and one site of disease that must be uni-dimensionally ≥ 10 mm considered as measurable according to RECIST v1.1. This lesion will not be treated by radiotherapy, however, note that lesion(s) that will be treated by radiotherapy will also be considered as measurable. Note that the largest size of the metastases to be irradiated will be 3cm and at that previous irradiation of these lesions is not allowed,
6. Life expectancy > 6 months,
7. At least one tumor site that can be biopsied for research purpose. Tumor lesion in close proximity to vascular structures such as large vessels, aneurysm or pulmonary arteriovenous malformation will not be considered for biopsy,
8. Availability of archived paraffin-embedded tumor tissue for research purpose,
9. Participant must have advanced disease and must not be a candidate for other approved therapeutic regimen known to provide significant clinical benefit based on investigator judgement,
10. Participants who received prior anti-PD-1/L1 therapy must fulfill the following requirements - population 3 and population 5 only

    * Have achieved a complete response, partial response or stable disease and subsequently had disease progression while still on anti-PD-1/L1 therapy
    * Have received at least two doses of an approved anti-PD-1/L1 therapy (by any regulatory authority)
    * Have demonstrated disease progression as defined by RECIST v1.1 within 18 weeks from the last dose of the anti- PD-1/L1 therapy.
11. Adequate hematological, renal, metabolic and hepatic functions
12. No prior or concurrent malignant disease needing an active treatment,
13. At least three weeks since last chemotherapy, immunotherapy or any other pharmacological treatment and/or radiotherapy,
14. Recovery to grade ≤ 1 from any adverse event (AE) derived from previous treatment, excluding alopecia of any grade and non-painful peripheral neuropathy grade ≤ 2,
15. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to inclusion.
16. Both women and men must agree to use an effective method of contraception throughout the treatment period and for five months after discontinuation of treatment.
17. Voluntary signed and dated written informed consents prior to any specific study procedure,
18. Participants with a social security in compliance with the French law.

Exclusion criteria:

1. Previous treatment with a TLR agonist
2. Evidence of progressive or symptomatic central nervous system (CNS) or leptomeningeal metastases,
3. Women who are pregnant or breast feeding,
4. Participation in a study involving a medical or therapeutic intervention in the last 30 days,
5. Known hypersensitivity to CHO cell products or to any involved study drug or of its formulation components,
6. History of severe allergic anaphylactic reactions to chimeric, human or humanized antibodies, or fusion proteins,
7. Treatment with systemic immunosuppressive medications including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF agents within 2 weeks prior to inclusion.
8. Major surgical procedure, open biopsy or significant traumatic injury within 28 days before inclusion,
9. Any of the following cardiac criteria: congestive heart failure ≥ New York Heart Association (NYHA) class 2, unstable angina, new-onset angina, myocardial infarction less than 6 months before inclusion, uncontrolled cardiac arrhythmias, known left ventricular ejection fraction (LVEF) <50%, previously experience of pericardial disorder
10. Individuals deprived of liberty or placed under legal guardianship,
11. Prior organ transplantation, including allogeneic stem cell transplantation,
12. Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis, cirrhosis, fatty liver and inherited liver disease,
13. History of intra-abdominal inflammatory process within the last 12 months such as, but not limited to, diverticulitis, peptic ulcer disease or colitis.
14. History of autoimmune disease including, but not limited to systemic lupus erythematosus (SLE), Sjögren's syndrome, glomerulonephritis, multiple sclerosis, rheumatoid arthritis, vasculitis, systemic immune activation, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Guillain-Barré syndrome, Bell's palsy.
15. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan.
16. Poorly controlled Type II diabetes mellitus defined as a screening fasting plasma glucose ≥160 mg/dL (or 8.8 mmol/L).
17. Severe infections within 2 weeks prior to inclusion, including but not limited to SARS-Cov-2 infection, hospitalization for complications of infection, bacteremia, or severe pneumonia.
18. Received therapeutic oral or IV antibiotics within 2 weeks prior to inclusion.
19. Participant has spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease is clinically stable at least 14 days prior to inclusion.
20. Administration of a live, attenuated vaccine within 4 weeks before the start of study medication .
21. Has known active hepatitis B or hepatitis C,known history of Human Immunodeficiency or known acquired immunodeficiency syndrome, known history of tuberculosis
22. Patients with current retinal disorder confirmed by retinal examination (external ocular examination, routine slit lamp biomicroscopy of anterior ocular structures and evaluation of the anterior and posterior chamber,
23. Patients who wear contact lenses unable to replace them with glasses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of the antitumor activity of atezolizumab combined with BDB001 and radiotherapy in patients with pancreatic cancer. | Within 6 months of treatment onset
  Antitumor activity will be assessed in terms of disease control rate within 24 weeks of treatment onset and is defined as the proportion of patients with complete response (CR), partial response (PR) or stable disease (SD) observed within 24 weeks of treatment onset (while treated with the investigational product), based on RECIST 1.1 criteria.
Assessment of the antitumor activity of atezolizumab combined with BDB001 and radiotherapy in patients with virus associated tumors. | Within 6 months of treatment onset
  Antitumor activity will be assessed in terms of disease control rate within 24 weeks of treatment onset and is defined as the proportion of patients with complete response (CR), partial response (PR) or stable disease (SD) observed within 24 weeks of treatment onset (while treated with the investigational product), based on RECIST 1.1 criteria.
Assessment of the antitumor activity of atezolizumab combined with BDB001 and radiotherapy in patients with non-small cell lung cancer. | Within 6 months of treatment onset
  Antitumor activity will be assessed in terms of disease control rate within 24 weeks of treatment onset and is defined as the proportion of patients with complete response (CR), partial response (PR) or stable disease (SD) observed within 24 weeks of treatment onset (while treated with the investigational product), based on RECIST 1.1 criteria.
Assessment of the antitumor activity of atezolizumab combined with BDB001 and radiotherapy in patients with soft-tissue sarcoma. | 6 months of treatment onset
  Antitumor activity will be assessed in terms of 6-month progression-free rat (PFR) and is defined as the proportion of patients with complete response (CR), partial response (PR) or stable disease (SD) observed at 6 months following treatment onset and more than 24 weeks, based on RECIST 1.1 criteria.
Assessment of the antitumor activity of atezolizumab combined with BDB001 and radiotherapy in patients with bladder cancer. | Within 6 months of treatment onset
  Antitumor activity will be assessed in terms of disease control rate within 24 weeks of treatment onset and is defined as the proportion of patients with complete response (CR), partial response (PR) or stable disease (SD) observed within 24 weeks of treatment onset (while treated with the investigational product), based on RECIST 1.1 criteria.
Assessment of the antitumor activity of atezolizumab combined with BDB001 and radiotherapy in patients with triple negative breast cancer. | Within 6 months of treatment onset
  Antitumor activity will be assessed in terms of disease control rate within 24 weeks of treatment onset and is defined as the proportion of patients with complete response (CR), partial response (PR) or stable disease (SD) observed within 24 weeks of treatment onset (while treated with the investigational product), based on RECIST 1.1 criteria.

SECONDARY OUTCOMES:
6-month Progression-free rate (PFR) in patients with pancreatic cancer. | 6 months
  Progression-free rate is defined as the rate of complete or partial response (CR, PR) or stable disease (SD), as per RECIST 1.1 criteria.
6-month Progression-free rate (PFR) in patients with virus-associated tumor. | 6 months
  Progression-free rate is defined as the rate of complete or partial response (CR, PR) or stable disease (SD), as per RECIST 1.1 criteria.
6-month Progression-free rate (PFR) in patients with non-small cell lung cancer. | 6 months
  Progression-free rate is defined as the rate of complete or partial response (CR, PR) or stable disease (SD), as per RECIST 1.1 criteria.
6-month Progression-free rate (PFR) in patients with bladder cancer. | 6 months
  Progression-free rate is defined as the rate of complete or partial response (CR, PR) or stable disease (SD), as per RECIST 1.1 criteria.
6-month Progression-free rate (PFR) in patients with triple negative breast cancer. | 6 months
  Progression-free rate is defined as the rate of complete or partial response (CR, PR) or stable disease (SD), as per RECIST 1.1 criteria.
6-month objective response rate (ORR) independently for each population. | 6 months
  Objective response is defined as the proportion of patients with complete response (CR) or partial response (PR) observed at 6 months, based on RECIST 1.1 criteria.
Objective response rate (ORR) within 24 weeks of treatment onset, independently for each population. | Within 6 months
  Objective response is defined as the proportion of patients with complete response (CR) or partial response (PR) observed within 24 wekks after treatment onset, based on RECIST 1.1 criteria.
Best overall response, independently for each population. | Throughout the treatment period, an expected average of 6 months
  Best overall response is defined as the best response across all time points (RECIST 1.1). The best overall response is determined once all the data for the patient is known (RECIST 1.1).
1-year progression-free survival, independently for each population. | 1 year
  Progression-free survival is defined as the delay between the start date of treatment and the date of progression (as per RECIST 1.1) or death (from any cause), whichever occurs first.
2-year progression-free survival, independently for each population. | 2 years
  Progression-free survival is defined as the delay between the start date of treatment and the date of progression (as per RECIST 1.1) or death (from any cause), whichever occurs first.
1-year overall survival, independently for each population. | 1 year
  Overall survival is defined as the delay between the start date of treatment and the date of death (of any cause).
2-year overall survival, independently for each population. | 2 years
  Overall survival is defined as the delay between the start date of treatment and the date of death (of any cause).
Safety profile, independently for each population: Common Terminology Criteria for Adverse Events version 5 | Throughout the treatment period, an expected average of 6 months
  Toxicity graded using the Common Terminology Criteria for Adverse Events version 5.
Tumor immune cells levels | before treatment onset and cycle 3 day 1 (each cycle is 21 days)
  Levels of immune cells in tumor will be measured by immunohistochemistry.
Blood cytokines levels | baseline, cycle 1 day 1, cycle 2 day 1, cycle 3 day 1 and progression (each cycle is 21 days)
  Levels of cytokines in blood will be measured by ELISA.
Blood lymphocytes levels | baseline, cycle 1 day 1, cycle 2 day 1, cycle 3 day 1 and progression (each cycle is 21 days)
  Levels of lymphocytes in blood will be measured by flow cytometry.
Blood kynurenine levels | baseline, cycle 1 day 1, cycle 2 day 1, cycle 3 day 1 and progression (each cycle is 21 days)
  Levels of kynurenine in blood will be measured by ELISA.

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - Institut Bergonié, Bordeaux
  - Chu Brest, Brest
  - Centre François Baclesse, Caen
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Hôpital La Timone, Marseille
  - Institut Paoli Calmettes, Marseille
  - Institut Curie, Paris
  - CHU Poitiers, Poitiers
  - Centre Eugène Marquis, Rennes
  - IUCT Oncopôle, Toulouse

IPD SHARING:
Plan to Share IPD: No